CLINICAL TRIAL: NCT01851707
Title: A Phase 2, Double-Blind, Parallel, Placebo-Controlled, Randomized Study to Evaluate Multiple Dose Levels of Duvelisib With Background Methotrexate in Subjects With Active Rheumatoid Arthritis and an Inadequate Response to Methotrexate Alone
Brief Title: A Double-Blind Study Evaluating Duvelisib in Subjects With Moderate to Severe Rheumatoid Arthritis and an Inadequate Response to Methotrexate Alone
Acronym: ASPIRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPI-145-04
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — duvelisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IPI-145, low dose BID (Experimental)
  Interventions: Drug: IPI-145
- IPI-145, medium dose BID (Experimental)
  Interventions: Drug: IPI-145
- IPI-145, high dose BID (Experimental)
  Interventions: Drug: IPI-145
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IPI-145 — 2 blinded capsules will be administered twice a day (morning and night) for 12 weeks.
  Arms: IPI-145, high dose BID; IPI-145, low dose BID; IPI-145, medium dose BID
Drug: Placebo — 2 blinded capsules will be administered twice a day (morning and night) for 12 weeks.
  Arms: Placebo BID

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of multiple dose levels of the investigational product (study drug), IPI-145, in combination with methotrexate compared to methotrexate alone in subjects with active moderate-to-severe Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This Phase 2 study is designed to examine the efficacy and safety of multiple dose levels of IPI-145 in subjects with active moderate-to-severe Rheumatoid Arthritis receiving a background stable dose of methotrexate. The study will employ a randomized, double-blind, placebo-controlled, parallel design.

Approximately 316 adult subjects who meet all eligibility criteria at Screening will be randomized at Baseline in a 1:1:1:1 ratio to one of 4 dose groups.

All treatments will be administered twice a day (BID). After randomization, subjects will enter a 12-week Treatment Period, where study drug (IPI-145 or placebo) will be self-administered BID as an outpatient. During the Treatment Period, subjects will return to the clinic for efficacy and safety assessments every 2 weeks. Following Treatment Period completion at Week 12, subjects will enter a 3-week Follow-up Period which includes one clinic visit approximately 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Rheumatoid Arthritis for at least 6 months
* Active disease, based on Screening clinical and laboratory criteria, despite taking methotrexate for at least 3 months

Exclusion Criteria:

* Pregnant or lactating females
* Previous failure or inadequate response to >2 biologic disease-modifying anti-rheumatic drugs (DMARDs)
* Concurrent DMARD treatment other than methotrexate, sulfasalazine, chloroquine, or hydroxychloroquine
* Treatment with > 10 mg daily prednisone (or equivalent) or more than one non-steroidal anti-inflammatory drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a 20% improvement in the American College of Rheumatology Criteria (ACR20) from Baseline to Week 12 | Baseline (Day 1), Weeks 2, 4, 6, 8, 10 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (64):
- Bulgaria (7):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
  - Targovishte
  - Varna
- Colombia (3):
  - Medellín, Antioquia
  - Bogota, Cundinamarca
  - Bucaramanga, Santander Department
- Germany (2):
  - Frankfurt
  - Halle
- Hungary (5):
  - Budapest
  - Kecskemét
  - Mezőkövesd
  - Nyíregyháza
  - Veszprém
- Mexico (10):
  - Mexico City, Col Roam Sur
  - Mexico City, Del Cuautemoc
  - León, Guanajuato
  - Guadalajara, Jalisco
  - Madero, Mexico DF
  - Morelia, Michoacán
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosi, C.P.
  - Mérida, Yucatán
  - Mexico City
- New Zealand (2):
  - Otahuhu, Auckland
  - Wellington
- Poland (13):
  - Grodzisk, Mazowiecki
  - Krakow, Okulickiego
  - Bialystok
  - Elblag
  - Krakow
  - Lublin
  - Nadarzyn
  - Poznan
  - Skierniewice
  - Sosnowiec
  - Stalowa Wola
  - Starachowice
  - Wroclaw
- Romania (5):
  - Baia Mare
  - Brăila
  - Bucharest
  - Oradea
  - Timișoara
- Russia (8):
  - Petrozavodsk, Republic of Karelia
  - Ryazan, Ryazan Oblast
  - Moscow
  - Orenburg
  - Saint Petersburg
  - Saratov
  - Vladimir
  - Yaroslavl
- Serbia (2):
  - Belgrade
  - Novi Sad
- Ukraine (7):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Poltava
  - Ternopil
  - Zaporizhzhya